CLINICAL TRIAL: NCT04251260
Title: Effectiveness of Positioning on the Movement and Clinical Physiological Outcomes of Preterm Neonates
Brief Title: Effectiveness of Positioning in Preterm Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Patras (Other)
Collaborators: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Theofani Bania, Assistant Professor, Department of Physiotherapy, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPatras2019
Record Dates: First submitted 2020-01-19; First posted 2020-01-31 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Premature Baby 26 to 32 Weeks; Preterm Birth
Keywords: preterm; positioning; snuggle up; general movements
MeSH Terms: conditions — Premature Birth | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the principal investigator who is not an assessor will know the allocation of the neonates to the 2 groups. The assessors will be blind to the allocation of the neonates.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positioning in flexion (Experimental): Intervention: Positioning of body in flexion and aligment towards midline with Snuggle up (Philips, USA)
  Interventions: Other: Positioning in flexion
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Positioning in flexion — The intervention group will be positioned in flexion (i.e. lower limbs in flexion, hand in midline) with an aid, the Snuggle up (Philips, USA). With positioning, the neonates bottom is tucked down in the snuggle up pocket, legs are aligned and gently flexed and hands towards midline and near the face.
  Positioning will be demonstrated to the nursing staff of the Neonatal Intensive Care Unit (NICU). The intervention group will receive positioning during day and night throughout the intervention period.
  Arms: Positioning in flexion

SUMMARY:
Introduction: When babies are born prematurely, they are deprived of their usual space limits (uterus walls). This along with the action of gravity to which they are exposed after birth, makes the neonates have a low muscle tone, acquire a posture of extension, being more irritable and having difficulties with their alertness-sleep cycle. There are few studies that have assessed the effectiveness of positioning of premature neonates. However, none of these studies has focused on exploring the effects of positioning on the patterns of movement and gross motor function of the pre-term neonates.

Aim: The aim of this study is to investigate the effects of positioning on the patterns of movement, gross motor development and physiological clinical outcomes of pre-term neonates.

Methods: A sample of pre-term neonates of ≤ 32 weeks of gestation from the Neonatal Intensive Care Unit (NICU) of the General University Hospital of Patras will be randomly assigned to two groups. The intervention group will receive positioning with Snuggle up (Philips, USA), while the control group will receive usual care. Outcomes will be assessed with the general movements of Prechtl and the Denver II scale at baseline and at term-age of each neonate. Physiological outcomes will be also assessed such as heart rate, respiratory rate, weight gained from baseline to term-age, days to achieve full oral feeding, days on the ventilator, days on oxygen, and duration of stay in the NICU. Basic characteristics of the neonates will be obtained from their medical record, i.e. weeks of gestation at birth, gender, type of birth (normal or Caesarian), weight at birth, and Αpgar score and will be used to compare the 2 groups for similarities at the baseline of the trial.

DETAILED DESCRIPTION:
Study Protocol

Introduction:

The NICU provides a sensory overload through excessive handling, noisy environment, neglected cry, prolonged sleep state and social interactions of the newborns with the professionals. All these make difficult the internal organization of the preterm neonate (Pereira et al, 2013). Also, when babies are born prematurely, their muscles have not yet acquired the appropriate tone which is normally low compared to the muscle tone of full-term neonates. With the deprivation of their usual space limits (uterus walls) and the action of gravity to which the neonates are exposed after birth, the preterm neonates acquire a posture of extension, which is contrary to the flexion they usually adopt in the uterus. This extension position does not help the flexion of their limbs and makes the hand-mouth activities and meeting the middle line difficult. Further, the deprivation of the physical rhythms of the neonates' usual space creates insecurity, irritability, increased extensive motor activity and difficulties with respiration and alertness-sleep cycle (Toso et al, 2015; Zarem et al, 2013).

There is a randomized controlled trial (RCT) that investigated the effectiveness of positioning on the general condition and ability to be fed of 100 neonates (≤ 32 weeks of gestation). This study compared a positioning using the Dandle Roo (DandleLion Medical) with traditional or other positioning (e.g. rolls of sheets, snuggle up) (Madlinger-Lewis et al, 2013). At term-age, a significant difference was found between the two groups, favoring the Dandle Roo positioning, in the movements symmetry as assessed with the NICU Network Neurobehavioral Scale (mean difference: 0.90, 95% confidence intervals: 0.05 to 1.75). No other significant differences were observed at rest of outcomes. Another RCT including 56 preterm neonates (27-32 weeks of gestation) explored the effects of positioning with the Snuggle up and Bendy Pumpers (Philips, USA) in comparison to traditional positioning (rolls of soft fabric). The results showed a significant difference between the two groups, favoring the intervention group, in respiratory rate, oxygen saturation, score of cardiovascular stability, and weight gain (p<0.5) (Sathish et al, 2017).

However, none of these previous studies has investigated any differences in the patterns of movement of the pre-term neonates after a positioning intervention. For example, no study has assessed the gross motor function of the pre-term neonates using the general movements of Prechtl after a positioning intervention, although this assessment is considered important for the prognosis of the motor development and ability for independence of these children (Einspieler et al, 2016). No previous study has also assessed the effect of positioning in the long-term neuro-developmental progress of pre-term children with scales such as the Denver II scale, which scale is also important for the prognosis of the development of the neonate.

Aim of the study:

The current trial aims at exploring the effectiveness of positioning in a "flexion" position on the movement and clinical outcome of neonates (≤32 weeks of gestation), which group of neonates is a high-risk group.

Methods:

Inclusion criteria: neonates of 32 weeks of gestation or less. Exclusion criteria: neonates with congenital deformities, genetic anomalies, or neurological deficits detected at 1st week post-natal, neonates of multiple birth (triplets and over) or breech deliveries.

Two groups of neonates will be randomly assigned using a concealed method (sealed envelopes) either to positioning (intervention group) or to usual care (control group). In order to maintain similar gestational ages throughout the two groups, participants will be stratified by gestational age (≤28 weeks and >28 weeks). Each stratum will have an independent randomization scheme.

The intervention group will be positioned in flexion (lower limbs in flexion, hands in midline) with a positioning aid, the Snuggle up (Philips, USA). With positioning, the neonates bottom is tucked down in the snuggle up pocket, legs are aligned and gently flexed and hands are placed towards midline and near the face. The control group will not receive any positioning in flexion and the neonates will lie as usually. This study has been approved by the Research Committee of the General University General Hospital of Patra (decision: 246, date: 09/04/2019).

Factors that may affect the neonates' condition should be controlled, and be similar to both groups of neonates. Such factors are light, noise, temperature of room (incubator), touching from nursing staff or others etc.

The intervention group will receive positioning during day and night throughout the intervention period. Neonates may be removed from positioning when a nurse or mother needs to feed them, that is a period that will not last more than 1 hour/day. The principal investigator (TB) will demonstrate the positioning to the Neonatal Intensive Care Unit (NICU) nursing staff, and will check each week during the intervention period the positioning of the neonates as well as will reply to any questions of the staff. The physiological status (normal functioning) of the neonates will be checked regularly by the neonatologist in charge and the nurses of the NICU.

Outcomes Assessments of the 2 groups (intervention and control group) will take place at baseline and again at term-age of each neonate. For assessment, the General Movements (GM's) of Prechtl (Einspieler et al, 2016) using 5-minute video observations of each neonate will be used. The GM's assessment is a non-invasive assessment and can be used from birth up to 5 months. In this study, the detailed GM's assessment will be conducted by two pediatric physiotherapists, independently. The two assessors have a long-lasting experience in assessing/treating small children and infants and will be blind to which group the neonates will be assigned. There is evidence that the GM's (total score) demonstrate high test-retest reliability with Intra-class Correlation Coefficients (ICCs) or Pearson coefficients exceeding 0.84 (Yeh et al, 2016), while there were lower correlation coefficients during the initial period of writhing movements (6-8 weeks post-natal). A significant amount of test-retest reliability was also found for each sub-category of the Detailed GM's assessment with ICCS exceeding 0.80, except for the assessment of "speed" (ICC: 0.51) (Yeh et al, 2016). Evidence of moderate to good intra-tester reliability has also been demonstrated (kappa coefficient: 0.44-0.63) (Bernhardt et al, 2011), and 97-100% agreement between raters for the GM's total score. Assessment will also be performed with the Denver II scale (at term-age and 4 months of corrected age). This scale has shown a significant amount of validity for assessing the neuro-developmental progress of babies and infants. The assessment with the Denver II scale will be performed by a neonatologist of the NICU, who will be blind to the neonates' assignment.

The principal investigator will film all the videos at baseline and at post-intervention (at term-age for each neonate). Video recording will follow a typical method of observation of the GM's, and each video will have a 5-minute duration for a more reliable observation of the movement of each neonate. Video recording will take place at least 30 minutes after the neonate is fed and during periods in which the neonate is awake and is moving. Other parameters that will be examined at baseline and post-intervention are the heart rate, respiratory rate, weight gained from baseline to post-intervention, days to achieve full oral feeding, days on the ventilator, days on oxygen, and duration of stay in the NICU. Demographics and basic characteristics of the neonates will be recorded such as weeks of gestation at birth, gender, type of birth (normal or Caesarian), weight at birth, and Αpgar score to compare the 2 groups for similarities at the baseline of the trial. These data will be obtained from the neonates' medical record.

Written information about the study will be provided to the neonates' parents and written consent will be asked from either the mother or father (or the guardian of the neonate) before the neonate enters the trial. Detailed information will be also provided to all the staff of the NICU involved in the study. A code number will be given to each neonate to maintain his/her anonymity, during data analysis and dissemination of results. Babies videos needed for assessment will not be accessible from internet or other sharing mediums.

Video recording The neonate will lie on his/her back in the incubator, with no clothes and dressed only with a diaper. The surface of the incubator should be flat and of plain color (e.g. white) with no patterns etc. to avoid interference with accurate scoring in movement assessment.

The neonate should be in a calm state, not irritated and not sleeping either. If the baby is crying and is unsettled it will be difficult to film, therefore, in this case the filming will be postponed and completed at an alternative time. It is best that the neonate cannot see the nurse or other person except for the person filming as this may attract the baby's attention. No dummies or toys should be used and no interaction with the neonate by talking or touching throughout the video recording period.

A simple camera on a tripod (height 1.5 meters), will be placed next to the incubator and above the neonate at an angle so that the neonate can be seen in the frame (including his/her feet and hands). As afore-mentioned, 5-minute videos will be recorded twice (at the beginning and at term-age).

Data analysis:

Data will initially be presented using mean and standard deviation (descriptive data). For comparisons between the intervention and control group, the ANOVA and independent t-test will be used (SPSS). Differences will be considered statistically significant when p value is <0.5.

ELIGIBILITY:
Inclusion Criteria:

* Νeonates of 33 weeks of gestation or less

Exclusion Criteria:

Νeonates

* with congenital deformities or genetic anomalies
* with neurological deficits detected at 1st week post-natal
* of multiple birth (triplets and over) or breech deliveries

Ages: 24 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline General movements at 40 weeks | From baseline to 40 weeks
  General Movements (GM's) of Prechtl using 5-minute video observations of each neonate for the assessment
Change from 40 weeks Denver II Developmental Screening Test at 4 months of corrected age | From 40 weeks to 4 months of corrected age
  The purpose of the test is to identify young children with developmental problems

SECONDARY OUTCOMES:
Change from baseline Beats per minute (heart rate ) at 40 weeks | From baseline to 40 weeks
  The heart rate will be measured with a monitor connected to the neonate
Change from baseline Breaths per minute (respiratory rate) at 40 weeks | From baseline to 40 weeks
  The respiratory rate will be measured with a monitor connected to the neonate
Change from baseline Weight at 40 weeks | From baseline to 40 weeks
  Weight gained during the intervention period measured with the NICU scales
Days till full feeding | Up to 40 weeks
  This information will be collected from each neonate's file
Days the neonate needed oxygen | Up to 40 weeks
  This information will be collected from neonates file
Duration of stay in the NICU | Up to 40 weeks
  This information will be collected from neonates file

CONTACTS AND LOCATIONS:
Overall Officials: Theofani Bania, Principal Investigator — University of Patras, Greece
Locations (1):
- University of Patras, Pátrai, Greece

REFERENCES:
- [Background] Toso BR, Viera CS, Valter JM, Delatore S, Barreto GM. Validation of newborn positioning protocol in Intensive Care Unit. Rev Bras Enferm. 2015 Nov-Dec;68(6):1147-53. doi: 10.1590/0034-7167.2015680621i. English, Portuguese. PMID 26676439
- [Background] Zarem C, Crapnell T, Tiltges L, Madlinger L, Reynolds L, Lukas K, Pineda R. Neonatal nurses' and therapists' perceptions of positioning for preterm infants in the neonatal intensive care unit. Neonatal Netw. 2013 Mar-Apr;32(2):110-6. doi: 10.1891/0730-0832.32.2.110. PMID 23477978
- [Background] Bernhardt I, Marbacher M, Hilfiker R, Radlinger L. Inter- and intra-observer agreement of Prechtl's method on the qualitative assessment of general movements in preterm, term and young infants. Early Hum Dev. 2011 Sep;87(9):633-9. doi: 10.1016/j.earlhumdev.2011.04.017. Epub 2011 May 26. PMID 21616611
- [Background] Sathish Y, Edward Lewis L, Angelitta Noronha J, George A, Snayak B, S Pai M, et al. Clinical Outcomes of Snuggle up Position Using Positioning Aids for Preterm (27-32 Weeks) Infants. Iranian Journal of Neonatology. 2017
- [Background] Pereira FL, Nogueira de Goes Fdos S, Fonseca LM, Scochi CG, Castral TC, Leite AM. [Handling of preterm infants in a neonatal intensive care unit]. Rev Esc Enferm USP. 2013 Dec;47(6):1272-8. doi: 10.1590/S0080-623420130000600003. Portuguese. PMID 24626374
- [Background] Madlinger-Lewis L, Reynolds L, Zarem C, Crapnell T, Inder T, Pineda R. The effects of alternative positioning on preterm infants in the neonatal intensive care unit: a randomized clinical trial. Res Dev Disabil. 2014 Feb;35(2):490-7. doi: 10.1016/j.ridd.2013.11.019. Epub 2013 Dec 25. PMID 24374602
- [Background] Einspieler C, Marschik PB, Pansy J, Scheuchenegger A, Krieber M, Yang H, Kornacka MK, Rowinska E, Soloveichick M, Bos AF. The general movement optimality score: a detailed assessment of general movements during preterm and term age. Dev Med Child Neurol. 2016 Apr;58(4):361-8. doi: 10.1111/dmcn.12923. Epub 2015 Sep 14. PMID 26365130
- [Background] Yeh KK, Liu WY, Wong AM, Chung CY, Lien R, Chuang YF. Intra-observer reliability of Prechtl's method for the qualitative assessment of general movements in Taiwanese infants. J Phys Ther Sci. 2016 May;28(5):1588-94. doi: 10.1589/jpts.28.1588. Epub 2016 May 31. PMID 27313378